CLINICAL TRIAL: NCT05701202
Title: Assessing the Impact of "Super-whey" vs. Isonitrogenous Whey on Muscle Protein Synthesis at Rest and in Response to Acute Resistance Exercise Across the Lifespan
Brief Title: Assessing the Impact of "Super-whey" vs. Isonitrogenous Whey on Muscle Protein Synthesis
Acronym: ARLA-WHEY
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nottingham (Other)
Responsible Party: Principal Investigator, Philip Atherton, Professor, University of Nottingham
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: ARLA-WHEY_PtA_CMMP
Record Dates: First submitted 2021-08-04; First posted 2023-01-27 (Actual); Last update posted 2023-01-27 (Actual); Status verified 2023-01

CONDITIONS: Sarcopenia
MeSH Terms: conditions — Sarcopenia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Super-Whey protein (Experimental): Both protein sources will be given in doses that are considered low/normal, both in relation to recommended dietary advice and commercially available supplements. As such, no adverse reactions or side effects are expected through consumption of these supplementations
  Interventions: Dietary Supplement: Super-Whey protein
- Isonitrogenous whey protein (Active Comparator): Both protein sources will be given in doses that are considered low/normal, both in relation to recommended dietary advice and commercially available supplements. As such, no adverse reactions or side effects are expected through consumption of these supplementations
  Interventions: Dietary Supplement: Isonitrogenous whey protein

INTERVENTIONS:
Dietary Supplement: Super-Whey protein — 2 different protein supplements (as above) will be given in a randomised crossover fashion to participants
  Arms: Super-Whey protein
Dietary Supplement: Isonitrogenous whey protein — 2 different protein supplements (as above) will be given in a randomised crossover fashion to participants
  Arms: Isonitrogenous whey protein

SUMMARY:
Skeletal muscle accounts for approximately 45-55% of total body mass in healthy adults and plays a pivotal role in whole-body metabolic health, locomotion and physical independence. Undesirable loss of skeletal muscle mass (atrophy) is, however, a common feature of many diseases and scenarios including ageing, bed rest/immobilisation, cancer and physical inactivity. Despite the exact mechanisms causing muscle atrophy being not yet fully understood, "anabolic resistance" (reduced muscle building in response to protein feeding and exercise) is thought to be key, especially for age-related skeletal muscle losses (known as sarcopenia). As such, the search for optimal strategies (e.g., exercise and/ or nutritional interventions) to combat this anabolic blunting remains a hot-topic in scientific research.

Leucine, an essential and branched chain amino acid (EAA/BCAA), is thought to be the most potent AA for stimulating muscle protein synthesis (MPS; the muscle building process). Although, as a stand-alone supplement, leucine is unlikely to provoke a robust and prolonged state of MPS, low doses of leucine-enriched mixed-EAAs can elicit similar increases in MPS as compared to a large dose of whey protein. As reduced appetite and increased satiety (feeling fuller) are common with advancing age, supplementation of a low-dose protein (i.e., leucine-enriched) that can adequately stimulate MPS may contribute to muscle health maintenance in older adults and reduce satiation following a meal.

This study aims to examine whether a novel whey protein with greater leucine content ("super-whey") has superior muscle building properties compared to a regular whey protein, at rest and after a single bout of exercise, in both young and older adults

ELIGIBILITY:
Inclusion Criteria:

* Participant is in the desired age-ranges (young adults: 18-35 years; older adults: 65+ years).
* Participant is willing and able to give informed consent for participation in the study.
* Participant is physically able to perform resistance exercise

Exclusion Criteria:

* A BMI <18 or >35 kg/m2
* Active cardiovascular, cerebrovascular or respiratory disease: e.g. uncontrolled hypertension (BP > 160/100), angina, heart failure (class III/IV), arrhythmia, right to left cardiac shunt, recent cardiac event, COPD, pulmonary hypertension or recent (6 mo) stroke
* Any metabolic disease
* Clotting dysfunction
* A history of, or current neurological or musculoskeletal conditions (e.g. epilepsy)
* Lactose intolerance
* Having taken part in a research study in the last 3 months involving invasive procedures or an inconvenience allowance

Ages: 18 Years to 85 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2021-06-15 (Actual); Primary Completion 2022-11-22 (Actual); Study Completion 2022-11-22 (Actual)

PRIMARY OUTCOMES:
Muscle protein fractional synthetic rate (postabsorptive) | Assessed at 3 hour mark
  Postabsorptive measures of muscle protein synthesis assessed in muscle tissue (collected by muscle biopsy). This outcome will be assessed prior to administering a protein drink to obtain muscle protein fractional synthetic rate in the fasted state.
Muscle protein fractional synthetic rate (postprandial) | Assessed at 6 hour mark
  Postprandial measures of muscle protein synthesis assessed in muscle tissue (collected by muscle biopsy). This outcome will be assessed following administering a protein drink to obtain muscle protein fractional synthetic rate in the fed state.

SECONDARY OUTCOMES:
Plasma amino acid concentrations | Assessed over 7.5 hours
  During the fasted and fed states of the study, blood samples are collected every 20 minutes to capture the plasma amino acid concentrations in the blood at that time-point (24 timepoints assessed). Future analysis using mass-spectroscopy will allow determination of the different amino acid concentrations in the blood plasma collected.

CONTACTS AND LOCATIONS:
Overall Officials: Philip Atherton, Prof, Principal Investigator — University of Nottingham
Locations (1):
- Centre of Ageing, Metabolism and Physiology, Derby, United Kingdom